CLINICAL TRIAL: NCT02523417
Title: HepaSphere Interventional Therapy Using Digital Subtraction Angiography（DSA for Breast Cancer: Clinical Trial
Brief Title: HepaSphere Interventional Therapy Using Digital Subtraction Angiography（DSA）for Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Breast Cancer HepaSphere
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2015-10

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; HepaSphere
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- HepaSphere (Experimental): breast cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）
  Interventions: Procedure: interventional therapy
- control (Placebo Comparator): breast cancer patients received traditional therapy
  Interventions: Procedure: interventional therapy

INTERVENTIONS:
Procedure: interventional therapy — breast cancer patients received HepaSphere interventional therapy using the digital subtraction angiography（DSA）

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of HepaSphere interventional therapy using digital subtraction angiography（DSA）for breast cancer.

DETAILED DESCRIPTION:
By enrolling patients with breast cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of HepaSphere interventional therapy using digital subtraction angiography（DSA）for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18-80
2. Karnofsky performance status >60
3. Diagnosis of breast cancer based on histology or the current accepted radiological measures.
4. Classification tumor,nodes,metastasis-classification(TNM) stage: Ⅱ,Ⅲ,Ⅳ
5. Will receive interventional therapy
6. Life expectancy: Greater than 3 months
7. Patients' routine blood test, liver function and kidney function have no obvious abnormalities
8. Ability to understand the study protocol and a willingness to sign a written informed consent document

Exclusion Criteria:

1. Patients with other primary tumor except breast cancer
2. History of coagulation disorders or anemia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-05; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse events | 1 year

SECONDARY OUTCOMES:
Percentage of lesions interventional therapy that show no sign of recurrence 12 months after | 1 year
Progress free disease (PFS) | 1 year
Overall survival (OS) | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Lizhi Niu, PhD, Study Chair — Fuda Cancer Hospital
Locations (1):
- Central laboratory in Fuda cancer hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Niu L, Chen J, Yao F, Zhou L, Zhang C, Wen W, Bi X, Hu Y, Piao X, Jiang F, Zeng J, Liu W, Li J, He L, Mu F, Zuo J, Xu K. Percutaneous cryoablation for stage IV lung cancer: a retrospective analysis. Cryobiology. 2013 Oct;67(2):151-5. doi: 10.1016/j.cryobiol.2013.06.005. Epub 2013 Jun 24. PMID 23806858
- See also: related information — http://www.ncbi.nlm.nih.gov/pubmed/25937772